CLINICAL TRIAL: NCT02358252
Title: Heart Rate Variability and Orthostatic Hypotension in Stroke Patients Evaluated by Intelligent Biosensor System
Status: Withdrawn | Type: Observational
Why Stopped: The device was under developed with some technical bugs.
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Other Study IDs: CCH-140103
Record Dates: First submitted 2015-01-28; First posted 2015-02-06 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Cerebrovascular Accident
Keywords: Heart Rate Variability; orthostatic hypotension; stroke; integrated intelligent biosensor system
MeSH Terms: conditions — Stroke; Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Orthostatic hypotension: Collection of information of body mass index, modified Ashworth scale, maximal voluntary contraction(MVC), heart rate variability(HRV).
  Tilt table test was used in this study to identify if the subjects with or without orthostatic hypotension.
- Non-orthostatic hypotension: Collection of information of body mass index, modified Ashworth scale, maximal voluntary contraction(MVC), heart rate variability(HRV) Tilt table test was used in this study to identify if the subjects with or without orthostatic hypotension.

SUMMARY:
This research investigated the heart rate variability (HRV) and stroke patients' orthostatic hypotension in hospitalized stroke patients accompanied with dizziness at varied tilting angle controlled by tilting table with intelligent biosensor.

DETAILED DESCRIPTION:
Stroke patients readily accompany with the occurrence of orthostatic hypotension. To earlier predict patients occurring dizziness during the tilt table test, this study utilized a self-developed integrated intelligent biosensor system to assist clinical staff efficiently and immediately assessing stroke patients with orthostatic hypotension. Further purposes were to survey the relationship between the orthostatic hypotension and heart rate variability (HRV) and find the predicted models of orthostatic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are first time to get stroke.

Exclusion Criteria:

* unstable physiological conditions, serious joint spasticity, use cortisol or calming drugs, other neurological diseases

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2019-12-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Change of Heart Rate Variability (HRV) | Baseline: before Tilt table test, resting position, measure HRV with 3 minutes interval, totally 7 HRVs were measured
  measure subject's HRV, every 3 mins during the Tilt table test

CONTACTS AND LOCATIONS:
Overall Officials: TaSen Wei, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan